CLINICAL TRIAL: NCT04116268
Title: The Effect of Obesity on Pregnancy and Fetal Outcome in Glucose Tolerant Mothers
Status: Completed | Type: Observational
Sponsor: University Malaysia Sarawak (Other)
Responsible Party: Principal Investigator, Dr Huai Heng, Loh, Associate Professor Dr., University Malaysia Sarawak
Other Study IDs: F05/SpGS/1548/2017
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity: BMI >23kg/m2
- Control: BMI 18-22.9kg/m2

SUMMARY:
The participants are divided into subjects or controls based on the BMI taken during the first trimester of pregnancy upon recruitment. Participants with a BMI of ≥23kg/m2 were recruited as subjects (labelled as obese group) and those with BMI of 18.5-23kg/m2 were recruited as controls. Total gestational weight gain was calculated based on the difference between third trimester weight and first trimester weight. All participants who fulfilled the inclusion and exclusion criteria were recruited after informed consent. Demographic data of all participants were recorded. At first trimester, the participants' weight and height were recorded for calculation of BMI. At every trimester visit, the following were recorded: i) blood pressure using sphygmomanometer after 15 minutes of rest ii) mid-stream urine for presence of proteinuria iii) weight. The participants were followed up until the point of delivery. Occurrence of adverse pregnancy outcome, fetal outcome, and birth weight were documented. The pregnancy outcomes measured in this study included the need of primary caesarian section, the occurrence of pregnancy-induced hypertension (PIH), pre-eclampsia, and gestational age at delivery. The neonatal outcomes measured in this study included neonatal intensive care unit (NICU) admission, stillbirth, preterm delivery, occurrence of macrosomia and low birth weight, and neonatal birth weight.

ELIGIBILITY:
Inclusion Criteria:

* First trimester of pregnancy
* Aged 18 years or older
* Able to come for follow up at least once per trimester

Exclusion Criteria:

* Underlying diabetes mellitus
* Gestational diabetes mellitus diagnosed via OGTT
* Known genetic disorders affecting growth at time of recruitment
* Known congenital anomalies at time of recruitment
* Conceived via artificial insemination
* Hepatitis B/C/HIV infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Pregnant during first trimester
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who develop pregnancy-induced hypertension | 9 months
Number of neonates who require neonatal intensive care unit admission | 9 months
Number of participants who develop pre-eclampsia | 9 months
Number of participants who require primary caesarian section | 9 months
Gestational age at delivery | 9 months
Number of stillbirth | 9 months
Number of preterm delivery | 9 months
Number of macrosomia at delivery | 9 months
  Birth weight more than 4000g
Number of low birth weight at delivery | 9 months
  Birth weight less than 2500g
Birth weight | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Huai Heng Loh, Principal Investigator — University Malaysia Sarawak
Locations (1):
- Universiti Malaysia Sarawak, Kuching, Sarawak, Malaysia